CLINICAL TRIAL: NCT04274842
Title: Dynamic Optical Coherence Tomography Imaging of Telangiectasia Prior to Intense Pulsed Light Treatment - an Opportunity to Target Treatment?
Brief Title: D-OCT of Facial Telangiectasia Treated With IPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Gregor Jemec, Professor, PhD, DmsC, Head of Dpt., Zealand University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SJ-651
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Telangiectasia
Keywords: Dynamic optical coherence tomography; facial telangiectasia; intense pulsed light; blood vessel dimensions; selective photothermolysis
MeSH Terms: conditions — Telangiectasis

STUDY DESIGN:
Intervention Model Description: prospective observational cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-OCT image observational (Other): Patients clinically eligible for IPL treatment of facial telangiectasia were D-OCT scanned before, after, 1-3 days after and 1 month after treatment
  Interventions: Other: observation by D-OCT

INTERVENTIONS:
Other: observation by D-OCT — observation by D-OCT before, after, 1-3 days after, and 1 month after IPL treatment

SUMMARY:
Objectives: To examine whether dynamic Optical Coherence Tomography (OCT) could characterize vessel dimensions and blood flow of telangiectasias before and after treatment with Intense Pulsed Light (IPL).

Methods: Dynamic-OCT (D-OCT) imaged telangiectasia characterized blood vessel width and depth, blood flow, and attenuation. Measurements were done immediately before and after, 1-3 days after, and 1 month after IPL treatment. Characterization of vessel dimensions at baseline were verified by a blinded observer. At one-month follow-up, clinical improvement was characterized as good, moderate or none and possible adverse effects were described.

DETAILED DESCRIPTION:
Introduction Telangiectasia of the face are a common facial cosmetic disorder and may cause severe psychological distress. Facial telangiectasia may be treated with pulsed dye laser (PDL) or intense pulsed light (IPL). Clinical results are not always satisfactory and numerous treatments may be necessary to achieve acceptable results. Unexperienced operators often depend on treatment guidelines provided by the manufacturer when selecting energy settings for treatment, while more experienced operators may be guided by the immediate post-treatment biological endpoints and history of adverse events from previous treatment sessions. Thus, several treatments are often needed to determine optimal energy settings for the individual patient.

In general, light energy must be targeted to individual blood vessel dimensions, when optimizing laser or IPL treatment of vascular lesions. In clinical practice it may however be challenging to decide vessel width, vessel depth and blood flow by merely looking at the skin.

Optical coherence tomography (OCT) is a non-invasive in vivo imaging technique, which provides images of superficial skin structures. It has previously been demonstrated that OCT can visualize facial telangiectasias before and after IPL treatment. Dynamic OCT (D-OCT) adds identification and measurement of superficial cutaneous blood vessels with great certainty. Therefore, the aim of this study was to investigate whether D-OCT could be utilized to characterize vessel dimensions and blood flow of facial telangiectasias before and after IPL treatment.

Material and Methods Patients with telangiectasias visiting the Department of Dermatology for IPL treatment of telangiectasia at the Zealand University Hospital, Roskilde, between February and November 2018 were offered participation after informed consent. The study was approved by the Science Ethics Committee of Region Zealand (Approval no.: SJ-651) and the Danish Data Protection Agency (Approval no.: REG-177-2017).

D-OCT imaging was done immediately before, 1-3 days after, and one month after scheduled IPL treatment. The D-OCT scans and IPL treatments were performed by two separate physicians and the treating physician was blinded to all information obtained by D-OCT.

The IPL treatments were performed using a Palomar ICONTM Laser and Intense Pulsed Light platform applying a MaxGTM Optimized Handpiece with a dual-band wavelength of 500-670 nm and 870-1200 nm.

Dynamic OCT scans were performed by the 1305 nm VivoSight DX (Michelson Diagnostics, Kent, UK) with penetration depth of approximately 1 mm and vertical/horizontal optical resolution of less than 5/7.5 µm, respectively.

Drawn templates of appropriate facial telangiectasia ensured consistency of consecutive scans. Measurements of vessel dimensions were performed at the most evident level at horizontal images and verified by a blinded observer (PLA). A blinded (PLA) as well as an un-blinded evaluator (EHT) characterized vascular morphology at horizontal images from baseline and one-month follow-up. Clinical observations at one-month follow-up included changes in facial telangiectasia and registration of any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* legally competent,
* at least 18 years of age
* persons able to read and understand spoken and written information in Danish or English.
* One or more facial telangiectasia

Exclusion Criteria:

* wounds or ulcers in area of facial telangiectasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
vessel width dimension | one-month follow-up
  measurement of vessel width on D-OCT images
vessel depth dimension | one-month follow-up
  measurement of vessel depth on D-OCT images
vessel blood flow | one-month follow-up
  measurement of vessel blood flow on D-OCT images
Attenuation | one-month follow-up
  measurement of attenuation on D-OCT images

OTHER OUTCOMES:
Relation of D-OCT detected vessel dimensions to clinical efficacy | one-month follow-up
  Clinical efficacy detected as good, moderate or none
Relation of D-OCT detected vessel dimensions to adverse effects | one-month follow-up
  Description of adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Gregor BE Jemec, DmSc, Prof., Principal Investigator — Zealand University Hospital - Roskilde
Locations (1):
- Zealand University Hospital Roskilde, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No